CLINICAL TRIAL: NCT00396942
Title: Evaluation of the Plasticity of the Primary Motor Cortex and Motor Learning in Parkinson's Disease
Brief Title: Motor Skill Learning in People With Parkinson's Disease
Status: Completed | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 070020; 07-N-0020
Record Dates: First submitted 2006-11-07; First posted 2006-11-08 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2008-10-03

CONDITIONS: Parkinson's Disease
Keywords: Electroencephalogram (EEG); Nerve Conduction Study; Transcranial Magnetic Stimulation (TMS); Motor Evoked Potential; Parkinson Disease; PD; Healthy Volunteer; HV
MeSH Terms: conditions — Parkinson Disease

SUMMARY:
This study will compare brain changes in people with Parkinson's disease with those of normal control subjects while they learn motor skills. People with Parkinson's disease sometimes have trouble learning new skills, but it is not known why. This study will use repetitive transcranial magnetic stimulation (rTMS), nerve conduction studies, and electroencephaolography (EEG) to look for differences in the way the brain changes with learning in people with Parkinson's disease.

Healthy normal volunteers and people with Parkinson's disease who are between 21 and 80 years of age may be eligible for this study. Participants undergo the following procedures in five visits to the NIH Clinical Center:

Visit 1

Medical and neurological examination.

Visit 2

Motor training. Participants perform a pinching movement once every other second, timed to a metronome, during rTMS. For TMS, a wire coil is held on the subject's scalp. A brief electrical current is passed through the coil, creating a magnetic pulse that stimulates the brain. The subject hears a click and may feel a pulling sensation on the skin under the coil. There may be a twitch in the muscles of the face, arm or leg. rTMS involves repeated magnetic pulses delivered in short bursts of impulses.

Visits 3 and 4

Brain physiology studies using rTMS, nerve conduction studies (electrical nerve stimulation) and EEG. A nerve at the subject's wrist is stimulated with electrical impulses to measure the speed with which nerves conduct electrical impulses and the strength of the connection between the nerve and the muscle. rTMS is performed for 20 minutes. The EEG measures the electrical activity of the brain (brain waves). For this test, electrodes (metal discs) are placed on the scalp with a conductive gel and the brain waves are recorded while the subject moves his or her thumb briskly for 20 minutes.

Visit 5

Subjects undergo rTMS for 20 minutes and have an EEG.

...

DETAILED DESCRIPTION:
Objective

The aims of the present study are to:

1. Clarify that the altered plasticity of the primary motor cortex (M1) in patients with Parkinson's disease (PD) is associated with impaired motor learning by using the paired associative stimulation (PAS) technique, which can enhance or inhibit the M1 excitability with paired stimulation to the contralateral peripheral nerve and cerebral cortex.
2. Elucidate that the altered plasticity of the M1 in patients with PD goes together with impaired sensorimotor integration via the basal ganglia-thalamocortical loop.

Study population

12 right-handed patients with PD

12 right-handed age-matched healthy volunteers

Design

Patients and age-matched healthy volunteers will complete five different sessions: Visit 1: clinical screening; Visit 2: motor learning session; Visit 3 and 4: the paired associative stimulation (PAS) sessions; Visit 5: the control session.

During the motor learning session, subjects will be asked to perform metronome-paced pinch of their index finger and thumb.

During the PAS sessions, they will receive 20 minutes of paired stimulation to the contralateral peripheral nerve stimulation and transcranial magnetic stimulation (TMS) at the appropriate timing for producing changes of the M1 excitability.

During the control session, they will receive 20 minutes of repetitive TMS without the peripheral nerve stimulation.

Outcome measures

For the motor learning session:

* peak acceleration (MPA) of thumb movement
* maximal peak force (MPF) between the index finger and thumb

For the PAS and control sessions:

* peak-to-peak motor evoked potential (MEP) amplitude
* resting motor threshold
* afferent inhibition
* event related desynchronization (ERD) and event related synchronization (ERS)

ELIGIBILITY:
* INCLUSION CRITERIA:
* Right-handed healthy volunteers (21-80 years old)
* Idiopathic PD confirmed by either the PI or an HMCS physician to establish the diagnosis and rule out any other neurologic condition that might affect cortical plasticity.
* Patients must fulfill categories 1 to 3 of the Modified Hoehn and Yahr Scale in the 'off-medication' state.

EXCLUSION CRITERIA:

* Subjects with a history of neurological disorder that might affect cortical plasticity including head injury with loss of consciousness and epilepsy, current use or a history of alcohol or drug abuse, psychiatric disorders requiring hospitalization, or prolonged treatment such as substance abuse addiction
* Subjects with dementia; mini mental state examination (MMSE) less than 25, frontal assessment battery (FAB) less than 13
* Subjects with other parkinsonian syndromes such as Lewy body disease, corticobasal degeneration, progressive supranuclear palsy, Binswanger disease and multiple system atrophy
* Subjects with marked tremor, dyskinesia or sensory disturbance
* Subject who have been treated with the subthalamic nucleus stimulation and pallidotomy
* Subjects who are unable to refrain from anti-parkinsonian medications for up to 15 hours on study days
* Subjects with significant hearing loss

The following exclusion criteria are due to the use of TMS:

* Subjects with cardiac pacemakers, intracardiac lines, implanted medication pump
* Subjects with blood vessel, cochlear, or eye implants
* Subjects with increased intracranial pressure as evaluated by clinical means
* Subjects with metal in the cranium
* Subjects with dental braces (but dental fillings are okay), metal fragments from occupational exposure or surgical clips in or near the brain

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24
Dates: Start 2006-11-02; Study Completion 2008-10-03

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Bliss TV, Lomo T. Long-lasting potentiation of synaptic transmission in the dentate area of the anaesthetized rabbit following stimulation of the perforant path. J Physiol. 1973 Jul;232(2):331-56. doi: 10.1113/jphysiol.1973.sp010273. PMID 4727084
- [Background] Buonomano DV, Merzenich MM. Cortical plasticity: from synapses to maps. Annu Rev Neurosci. 1998;21:149-86. doi: 10.1146/annurev.neuro.21.1.149. PMID 9530495
- [Background] Dan Y, Poo MM. Spike timing-dependent plasticity of neural circuits. Neuron. 2004 Sep 30;44(1):23-30. doi: 10.1016/j.neuron.2004.09.007. PMID 15450157